CLINICAL TRIAL: NCT05074836
Title: Effects of Yili Child Formula Milk on Bone Health in 4-6 Year Children: a 12-month Randomized Controlled Trial
Brief Title: Milk Supplementation and Bone Health in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Collaborators: LanZhou University (Other)
Responsible Party: Principal Investigator, Yu-ming Chen, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SYSU-51000-20210723-0001
Record Dates: First submitted 2021-09-10; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Bone Density Increased; Body Height
Keywords: milk; bone health; body growth; young children
MeSH Terms: conditions — Osteosclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The two milk products have the same-looking package and similar taste.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Formula Milk (Experimental): Formula milk designed for young children aged over 3 years;
  Dosage: 195 ml/time;
  Frequence: 2 times /day;
  Duration: 12 months
  Interventions: Dietary Supplement: Formula milk
- Regular milk (Active Comparator): Regular milk (pure milk);
  Dosage: 195 ml/time;
  Frequence: 2 times /day;
  Duration: 12 months
  Interventions: Dietary Supplement: Regular milk
- Control foods (Other): Grain foods: e.g., bread;
  Dosage: 20-40 g/time;
  Frequence: 2 times /day;
  Duration: 12 months
  Interventions: Other: Control foods

INTERVENTIONS:
Dietary Supplement: Formula milk — Brand name: Yili (QQ star formula milk);
  Type: SCI-PRO NUTRI 5+6TM formula milk designed for young children aged over 3 years;
  Dosage: 195ml*2/d;
  Intervention duration: 12 months
  Arms: Formula Milk
Dietary Supplement: Regular milk — Brand name: Yili；
  Type: regular milk (pure milk);
  Dosage: 195ml*2/d;
  Intervention duration: 12 months
  Arms: Regular milk
Other: Control foods — Brand: N/A;
  Food type: grain foods (e.g., bread);
  Dosage: 20-40g * 2/d grain foods
  Intervention duration: 12 months
  Arms: Control foods

SUMMARY:
Objectives: to examine the effects of a Yili child formula milk and regular milk on bone health and growth in young children.

Study design: cluster randomized controlled trial.

Setting: kindergartens in Hui-ning County of Gansu Province, China (north west).

Participants: >=246 apparent healthy children aged 4-6 years old.

Interventions:

(I) Yili child formula milk (QQ star formula, SCI-PRO NUTR5+6TM), 195 ml *2 /day; (II) Yili regular milk (pure milk), 195ml*2 /day; (III) Controls: about 50g/d grain foods (containing 20-30 g carbohydrates), e.g. bread.

Interventional Duration: 12 months.

Outcome measures: determined at 0, 6 and 12 months post treatments. Primary outcomes: bone density and bone mineral contents at the forearm and heel, bone biomarkers.

Secondary outcomes: (1) anthropometric indices: weight, height, waist circumference, etc.; (2) immune status.

Other measures: dietary intakes, physical activities, general information, medical information, adverse of side effects.

Data Analyses: The one-year changes and percent changes in the primary and secondary outcomes will be compared among the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 4-6 years;
* female and male
* Can be enrolled into kindergarten/school as a normal child.
* Be willing to drinking milk daily.

Exclusion Criteria:

* Milk allergy or intolerance, did not to be used to drinking milk;
* Had the following diseases/conditions confirmed by a hospital: serious diseases of heart, liver, kidney, brain, hematopoietic system, immunity, thyroid or cancer that need to be hospitalization for more than 1 week or take medication(s) for more than 1 month with the past two years.
* having infectious diseases, e.g., tuberculosis, hepatitis, etc.
* Taking vitamin D, calcium tables or nutrient package;
* Consumed more than 3 times (>600ml) milk each week in the previous month.
* Be not willing to provide informed consent, or have other conditions that were considered to be unsuitable for the study by the investigators.
* Increases of body health were out of the range between 5-8 cm in the last year.

Ages: 48 Months to 83 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 254 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline bone mineral density (BMD) at 12 months | 0 and 12 months
  BMD (g/cm2) determined by a dual energy x-ray absorptiometry (DXA) at the left forearm and heel
Change from baseline bone mineral density (BMD) at 6 months | 0 and 6 months
  BMD (g/cm2) determined by DXA at the left forearm and heel
Change from baseline bone mineral contents (BMC) at 12 months | 0 and 12 months
  BMC (g) determined by DXA at the left forearm and heel.
Change from baseline bone mineral contents (BMC) at 6 months | 0 and 6 months
  BMC (g) determined by DXA at the left forearm and heel.
Change from baseline of bone-specific alkaline phosphatase at 12 months | 0 and 12 months
  Bone turnover marker 1: Bone-specific alkaline phosphatase
Change from baseline of bone-specific alkaline phosphatase at 6 months | 0 and 6 months
  Bone turnover marker 1: Bone-specific alkaline phosphatase
Change from baseline of osteocalcin at 12 months | 0 and 12 months
  Bone turnover marker 2: osteocalcin
Change from baseline of osteocalcin at 6 months | 0 and 6 months
  Bone turnover marker 2: osteocalcin
Change from baseline of C-terminal telopeptide of type I collagen at 12 months | 0 and 12 months
  Bone turnover marker 3: C-terminal telopeptide of type I collagen
Change from baseline of C-terminal telopeptide of type I collagen at 6 months | 0 and 6 months
  Bone turnover marker 3: C-terminal telopeptide of type I collagen
Change from baseline of tartrate resistant acid phosphatase at 12 months | 0 and 12 months
  Bone turnover marker 4: tartrate resistant acid phosphatase
Change from baseline of tartrate resistant acid phosphatase at 6 months | 0 and 6 months
  Bone turnover marker 4: tartrate resistant acid phosphatase

SECONDARY OUTCOMES:
Change from baseline body weight at 12 months | 0 and 12 months
  Anthropometric indices: body weight
Change from baseline body height at 12 months | 0 and 12 months
  Anthropometric indices: body height
Change from baseline biomarker of body growth at 12 months | 0 and 12 months
  Biomarker of body growth: insulin-like growth factor 1
Change from baseline immune globulin M (Ig M）at 12 months | 0 and 12 months
  Immune status: Blood Ig M
Change from baseline immune globulin G (Ig G）at 12 months | 0 and 12 months
  Immune status: Blood Ig G
Change from baseline immune globulin G (Ig A）at 12 months | 0 and 12 months
  Immune status: Blood Ig A
Change from baseline whit blood cell at 12 months | 0 and 12 months
  Immune status: whit blood cell

OTHER OUTCOMES:
Concentrations of blood total 25-hydroxide-vitamin D (25-OH-VD) | 0, 6 and 12 months
  Serum 25-OH-VD
Concentrations of blood parathyroid Hormone (PTH) | 0, 6 and 12 months
  Serum PTH
Nutritional status 1: Body weight | 0, 4, 8 and 12 months
  Body weight (in kg)
Nutritional status 2: waist circumference | 0, 4, 8 and 12 months
  Waist circumference (in cm)
Nutritional status 3: middle-arm circumference | 0, 4, 8 and 12 months
  Middle-arm circumference (in cm)
Nutritional status 4: skinfold thickness | 0, 4, 8 and 12 months
  Skinfold thickness (in mm)
Total consumption of milk and dairy food | 0, 4, 8 and 12 months
  Total consumption of milk and dairy food (in ml/d)
Consumption of dietary energy | 0, 4, 8 and 12 months
  Consumption of dietary energy (in kcal/d)
Consumption of dietary protein | 0, 4, 8 and 12 months
  Consumption of dietary protein (in g/d)
Consumption of dietary calcium | 0, 4, 8 and 12 months
  Consumption of dietary calcium (in mg/d)
Number of participants with treatment-related adverse events | 0, 4, 8 and 12 months
  Adverse events : assessed by using questionnaires of medical conditions, medications related to milk intake
Child behaviors | 0 and 12 months
  Child behaviours: assessed by using a Child behavior Questionnaire-- parent version. The minimum and maximum values: 26-78; higher scores mean worse outcome.
Physical activity | 0, 4, 8 and 12 months
  Physical activity (in MET, h/week): assessed by a Child Physical Activity Questionnaire
Concentrations of serum calcium | 0, 6 and 12 months
  Serum calcium (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Chen, Ph.D., Principal Investigator — Sun Yat-sen University; Zhifu Zhao, M. Phil, Study Chair — Inner Mongolia Dairy Technology Research Institute Co., Ltd.
Locations (1):
- Lanzhou University, Lanzhou, Gangshu, China

IPD SHARING:
Plan to Share IPD: No
Published data based on reasonable request.

REFERENCES:
- [Derived] Zhao ZF, Li BY, He Q, Hao JY, Zhang KS, Zhang B, Hu W, Feng HT, Szeto IM, Chen YM, Zhang GX, Tang XY. Impact of dairy supplementation on bone acquisition in children's limbs: a 12-month cluster-randomized controlled trial and meta-analysis. Arch Osteoporos. 2024 Jul 24;19(1):65. doi: 10.1007/s11657-024-01422-2. PMID 39043915